CLINICAL TRIAL: NCT01698294
Title: A Pilot Study of the Flaxseed Effects on Hormones and Lignans: Role of Race, Genes, and Gut Microbiome
Brief Title: Biomarkers in Post-Menopausal Women Receiving Flaxseed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); National Cancer Institute (NCI) (NIH); State University of New York at Buffalo (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: I 216812; NCI-2012-01246 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 216812 (Other: Roswell Park Cancer Institute); U01CA161809 (NIH)
Record Dates: First submitted 2012-09-04; First posted 2012-10-02 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: No Evidence of Disease
Keywords: gut microbiome; hormones; women; race; phytoestrogens
MeSH Terms: interventions — Watchful Waiting; Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (flaxseed) (Experimental): Participants receive flaxseed PO daily for 6 weeks. After a usual diet "washout" period of 8 weeks, patients crossover to Group II.
  Interventions: Dietary Supplement: Flaxseed; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Group II (usual diet) (Active Comparator): Participants maintain a usual diet for 6 weeks. After a usual diet "washout" period of 8 weeks, patients crossover to Group I.
  Interventions: Other: Clinical Observation; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Clinical Observation — Participants maintain usual diet and undergo clinical observation
  Arms: Group II (usual diet)
Dietary Supplement: Flaxseed — Given PO
  Other Names: FLAX SEED; Flour, Flaxseed; Linseed
  Arms: Group I (flaxseed)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies biomarkers in post-menopausal women receiving flaxseed. Studying samples of blood, urine, and feces in the laboratory from participants receiving flaxseed may help doctors understand the effects of flaxseed on biomarkers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine associations between the composition of the gut bacterial communities and baseline levels of the mammalian lignans and steroid hormones.

II. To determine how variation in gut microbial community composition and in steroid hormone and xenobiotic metabolizing genes affects the metabolism of mammalian lignans and steroid hormones after exposure to a lignan-rich food (flaxseed).

III. To determine how these associations differ by race (i.e., African American and European American women).

OUTLINE: Participants are randomized to 1 of 2 treatment groups.

GROUP I: Participants receive flaxseed orally (PO) daily for 6 weeks. After a usual diet "washout" period of 8 weeks, patients crossover to Group II.

GROUP II: Participants maintain a usual diet for 6 weeks. After a usual diet "washout" period of 8 weeks, patients crossover to Group I.

After completion of study treatment, participants are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Participant must be a non-Hispanic white or non-Hispanic black (self-reported race) woman 45 to 80 years of age and postmenopausal; postmenopausal will be defined as no menstrual cycle in the past 12 months; women with a hysterectomy but with intact ovaries will be included if aged >= 55 years
* Willingness to comply with the requirements of the study

Exclusion Criteria:

* Unwilling or unable to follow protocol requirements
* Self-reported race other than non-Hispanic white or non-Hispanic black
* Use, in the 2 months prior to week 1 visit, of antibiotics, hormone replacement therapy, nonprescription hormones or herbal supplements for menopausal symptoms, or flaxseed supplements
* Nut or seed allergy
* Self-reported inflammatory bowel disease
* Gastric bypass
* Use of thyroid replacement medication (Synthroid or similar) for < 1 year
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive flaxseed
* Chemotherapy/radiation within the past year
* Body weight greater than 400 pounds (limit of Tanita scale)

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Relative percent of Eubacteria composition from quantitative polymerase chain reaction (qPCR) associated with lignan levels | Up to week 21
Steroid hormone and lignans levels after exposure to a lignan-rich food (flaxseed) | Up to week 21

CONTACTS AND LOCATIONS:
Overall Officials: Spencer Rosario, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] McCann SE, Rodriguez EM, Erwin D, Yao S, Tritchler D, Hullar MAJ, O'Connor T, Lampe JW. Recruitment and Retention of Healthy, Postmenopausal Women of African and European Ancestry: Results from a Dietary Intervention with Repeated Biospecimen Collections. Curr Dev Nutr. 2022 Jan 29;6(3):nzac012. doi: 10.1093/cdn/nzac012. eCollection 2022 Mar. PMID 35261959